CLINICAL TRIAL: NCT01520415
Title: A Prospective, Randomized, Double-blind, Clinical Trial of Trigger Point Injection Therapy for the Treatment of Myofascial Pain Syndrome
Brief Title: Clinical Trial Examining the Short and Long-term Effect of Myofascial Trigger Points Injection in Low Back Pain Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Yoram Shir (Other)
Responsible Party: Sponsor-Investigator, Dr. Yoram Shir, Doctor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AEPMU-01
Record Dates: First submitted 2012-01-11; First posted 2012-01-30 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Bupivacaine; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupivacaine (Active Comparator)
  Interventions: Drug: Bupivacaine
- saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine — 2ml per injection up to a maximum of 8ml (4 identified trigger points) per visit
  Other Names: lidocaine
  Arms: bupivacaine
Drug: Saline — 2ml per injection up to a maximum of 8ml (4 identified trigger points) per visit
  Arms: saline

SUMMARY:
The objective of this study is to examine the short and long-term effect of myofascial trigger point injections with either a local anesthetic or saline in patients with chronic low back pain presenting with myofasical pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* CLBP of non-malignant origin, with or without accompanying leg pain, including patients with history of previous back surgery or trauma
* MPS as evident by at least one active MTP, located medial or lateral to the posterior iliac crest involving the gluteus maximus or medius, quadratus lumborum and erector spinae muscles
* While not precluding the participation in the study, MTP in other areas will not make patients eligible
* Pain lasting for at least six months

Exclusion Criteria:

* Any current motor weakness, but not sensory loss or abnormal reflexes in the lower limbs
* Any injection or nerve block in the low back in the last 6 months
* Local or systemic infection
* Bleeding disorder or the use of anticoagulation medications
* Known allergy to local anesthetics
* Poor understanding of written and spoken English or French

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold of the myofascial trigger points | 12 weeks
  Change in the pressure pain threshold will be measured using a pressure algometer.

SECONDARY OUTCOMES:
Pressure pain threshold of MTPs | baseline, 4 weeks, 8 weeks
  Change in the pressure pain threshold of MTPs after each MTP injection.
VAS Low Back Pain | baseline, 4 weeks, 8 weeks, 12 weeks
  Change in pain intensity after each MTPI and at the end of the study.
Roland-Morris Disability Questionnaire (RDQ-20) | baseline, 4 weeks, 8 weeks, 12 weeks
  Change in disability levels after each MTPI and at the end of the study.
Short-Form Health Status Survey 12 (SF-12) | baseline, 4 weeks, 8 weeks, 12 weeks
  Change in functional status, well-being and quality of life after each MTPI and at the end of the study.
Consumption of analgesic medications | 12 weeks
  Change in the consumption of analgesic medications.
Number of participants with Adverse Events | 12 weeks
  Adverse events resulting from the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Shir, MD, Principal Investigator — MUHC-RI
Locations (1):
- Alan Edwards Pain Management Unit - Montreal General Hospital, Montreal, Quebec, Canada